CLINICAL TRIAL: NCT02397135
Title: Control Ovarian Stimulation Timing Test
Acronym: COST2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-102
Record Dates: First submitted 2015-03-05; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Infertility
Keywords: genomic markers
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Granulosa cells as aspirated from the pre-ovulatory follicles
Oversight: Data Monitoring Committee: No

SUMMARY:
IVF (in vitro fertilization) cycles fails more often than they succeed. Surprisingly very little effort is invested in defining the reasons for failure and possibly finding ways to improve the success on the next cycle. The investigators believe that the main reasons for failure are related to oocyte quality and indirectly to the follicle response for a particular patient. The investigators have developed a panel of biomarkers to assess the faulty follicular conditions leading to lower oocyte quality. Using these markers would indicate if a given cycle was characterized by over growth, over-luteinization, early or late trigger. Indeed our transcriptomics analysis has identified biomarkers of follicles still in their growth phase at trigger or follicles that have already begun luteinisation compare to follicle that are at the optimal level of differentiation. Measuring these biomarkers would allow making a better diagnostic for a given patient and potentially explaining reasons for failure. The system would also become adjustable to variable COS (control ovarian stimulation) and individual clinical practices. It is important to realize that this is applicable to almost all cycle failure and can be done on a pool of follicular cells when none of the oocytes obtained has led to a pregnancy. This does not resolve uterine problems but often these are caused by hormonal conditions established by the ovary or the ovarian treatment. This technology can be applied in all IVF clinics as no special equipment is required. It would be particularly valuable in clinics where a number of cycles is limited due to funding, or in clinic where a package of 3 cycles is proposed to the patient. The patient interest to have a custom treatment increases at each failing cycle as well as the doctors' interest to succeed. This technology is not clinically validated yet and would require a period of testing where participating clinics will collect the samples for a retrospective analysis (presence of biomarkers of follicular problems vs outcome) then in a prospective analysis where the diagnostic is used in a sub-set of patient to modulate the second/third cycle compared the outcome to patient with no diagnostic. The increase in pregnancy rate or cumulative pregnancy rate should reach a minimum of 10 and 25 % respectively to indicate a significant value.

DETAILED DESCRIPTION:
IVF (in vitro fertilization) cycles fails more often than they succeed. Surprisingly very little effort is invested in defining the reasons for failure and possibly finding ways to improve the success on the next cycle. We believe that the main reasons for failure are related to oocyte quality and indirectly to the follicle response for a particular patient. We have developed a panel of biomarkers to assess the faulty follicular conditions leading to lower oocyte quality. Using these markers would indicate if a given cycle was characterized by over growth, over-luteinization, early or late trigger. Indeed our transcriptomics analysis has identified biomarkers of follicles still in their growth phase at trigger or follicles that have already begun luteinisation compare to follicle that are at the optimal level of differentiation. Measuring these biomarkers would allow making a better diagnostic for a given patient and potentially explaining reasons for failure. The system would also become adjustable to variable COS (control ovarian stimulation) and individual clinical practices. It is important to realize that this is applicable to almost all cycle failure and can be done on a pool of follicular cells when none of the oocytes obtained has led to a pregnancy. This does not resolve uterine problems but often these are caused by hormonal conditions established by the ovary or the ovarian treatment.

This technology can be applied in all IVF clinics as no special equipment is required. It would be particularly valuable in clinics where a number of cycles is limited due to funding, or in clinic where a package of 3 cycles is proposed to the patient. The patient interest to have a custom treatment increases at each failing cycle as well as the doctors' interest to succeed.

This technology is not clinically validated yet and would require a period of testing where participating clinics will collect the samples for a retrospective analysis (presence of biomarkers of follicular problems vs outcome).

Five Canadian IVF clinics have agreed to provide a minimum of 200 anonymized samples with information on the cycle/patient medical status. From these samples, RNA will be extracted and the gene expression level will be measured for 3 housekeeping genes and 21 markers derived from previous studies (Hamel et al 2008 and 2010, Nivet et al 2015 submitted).

The genes leading to the best predictive value of negative outcome will then be classified according to our understanding of ovarian physiology as key indicator for generating a diagnostic. The read-outs provided to the clinic would then be one of the 5 following: Too early trigger, too late trigger, too high stimulation (FSH), too high differentiation (LH) or time spread response (a combination of immature and over mature follicles)

ELIGIBILITY:
Inclusion Criteria:

* female Infertility

Exclusion Criteria:

* PCO (polycystic ovary) syndrome women over 42 male factor resulting in sperm samples less than 5 millions motile.

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: IVF (In vitro fertilisation) patients infertile patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Changes in gene expression levels between pregnant and non pregnant patients (ratio over housekeeping n=3) using 21 biomarkers to assess ovarian stimulation successes. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Andre Sirard, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

REFERENCES:
- [Background] Hamel M, Dufort I, Robert C, Gravel C, Leveille MC, Leader A, Sirard MA. Identification of differentially expressed markers in human follicular cells associated with competent oocytes. Hum Reprod. 2008 May;23(5):1118-27. doi: 10.1093/humrep/den048. Epub 2008 Feb 28. PMID 18310048
- [Background] Hamel M, Dufort I, Robert C, Leveille MC, Leader A, Sirard MA. Genomic assessment of follicular marker genes as pregnancy predictors for human IVF. Mol Hum Reprod. 2010 Feb;16(2):87-96. doi: 10.1093/molehr/gap079. Epub 2009 Sep 24. PMID 19778949
- [Background] Hamel M, Dufort I, Robert C, Leveille MC, Leader A, Sirard MA. Identification of follicular marker genes as pregnancy predictors for human IVF: new evidence for the involvement of luteinization process. Mol Hum Reprod. 2010 Aug;16(8):548-56. doi: 10.1093/molehr/gaq051. Epub 2010 Jul 7. PMID 20610614